CLINICAL TRIAL: NCT00951652
Title: Cognitive and Interpersonal Therapies for Generalized Anxiety
Brief Title: Efficacy of Adding Interpersonal and Emotional Processing Therapy Techniques to Cognitive Behavioral Therapy to Treat Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle G. Newman (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Michelle G. Newman, Study Director, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH058593-02 (NIH); R01MH058593-02 (NIH)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Generalized Anxiety Disorder
Keywords: CBT; GAD; Interpersonal Therapy; Emotion-Focused Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- CBT plus supportive listening (Experimental): 14 weekly therapy sessions, the first hour of which will be devoted to standard CBT techniques and the second hour will be supportive listening
  Interventions: Behavioral: CBT; Behavioral: supportive listening
- CBT plus Interpersonal and emotional processing therapy (Active Comparator): 14 weekly therapy sessions, the first hour of which will be devoted to standard CBT techniques and the second hour will be Interpersonal and emotional processing therapy
  Interventions: Behavioral: CBT; Other: Interpersonal and emotional processing therapy

INTERVENTIONS:
Behavioral: CBT
Other: Interpersonal and emotional processing therapy
  Arms: CBT plus Interpersonal and emotional processing therapy
Behavioral: supportive listening
  Arms: CBT plus supportive listening

SUMMARY:
This study will test a version of cognitive behavioral therapy for generalized anxiety disorders that incorporates interpersonal and emotional processing techniques.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is characterized by chronic worry that interrupts normal functioning. Some research has shown cognitive behavioral therapy (CBT) to be an effective treatment for GAD, but only half of people treated with CBT for GAD experience treatment benefits long-term. Standard CBT for GAD may lose effectiveness over time because it does not address interpersonal and emotional processing problems. This study will determine the efficacy of a version of CBT with additional therapeutic techniques for addressing interpersonal interactions and emotional processing among adults with GAD.

Participation in this study will include 14 weeks of treatment and 2 years of follow-up visits. All participants will receive 14 weekly, 2-hour, individual therapy sessions and one maintenance session scheduled after completing treatment. During the first hour of each session, all participants will receive standard CBT. Participants will be randomly assigned to receive one of two therapies during the second hour: training in interpersonal and emotional processing techniques or listening therapy. Participants may continue taking their current medications if they maintain a fixed dosage and keep a daily dairy of medication use, starting 2 weeks before study entry and lasting throughout treatment.

In-depth study assessments will take place at baseline and after completing the 14 weeks of therapy. Assessments will include clinical interviews, self-report questionnaires, and a physiological measurement session. Questions will pertain to anxiety symptoms, self-perceptions, emotional experience, and perceptions of the world. The physiological measurement session will involve recording bodily reactions, including brain waves, heart rate, eye movement, and breathing, while performing simple perceptual tasks. Brief psychological assessments will also follow each therapy session. Follow-up assessments conducted 6, 12, and 24 months after completing treatment will involve interviews and questionnaires as well as recording a week's worth of medication diaries.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of generalized anxiety disorder (GAD), as defined by the DSM-IV and agreed on by two diagnostic interviewers
* Clinician's Severity Rating for GAD of 4 (moderate) or greater

Exclusion Criteria:

* Concurrent psychosocial therapy or past adequate dosage of CBT
* Any medical contributions to anxiety
* Current substance abuse, psychosis, or organic brain syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 1998-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | Measured at baseline, post-treatment, and at 6-, 12-, and 24-month follow-ups
  Anxiety measures

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Newman, PhD, Study Director — Penn State University; Thomas D. Borkovec, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Newman MG, Llera SJ. A novel theory of experiential avoidance in generalized anxiety disorder: a review and synthesis of research supporting a contrast avoidance model of worry. Clin Psychol Rev. 2011 Apr;31(3):371-82. doi: 10.1016/j.cpr.2011.01.008. Epub 2011 Jan 26. PMID 21334285
- [Background] Newman MG, Castonguay LG, Borkovec TD, Fisher AJ, Boswell JF, Szkodny LE, Nordberg SS. A randomized controlled trial of cognitive-behavioral therapy for generalized anxiety disorder with integrated techniques from emotion-focused and interpersonal therapies. J Consult Clin Psychol. 2011 Apr;79(2):171-81. doi: 10.1037/a0022489. PMID 21443321
- [Background] Przeworski A, Newman MG, Pincus AL, Kasoff MB, Yamasaki AS, Castonguay LG, Berlin KS. Interpersonal pathoplasticity in individuals with generalized anxiety disorder. J Abnorm Psychol. 2011 May;120(2):286-98. doi: 10.1037/a0023334. PMID 21553942
- [Result] Boswell JF, Llera S, Newman MG, Castonguay LG. A Case of Premature Termination in a Treatment for Generalized Anxiety Disorder. Cogn Behav Pract. 2011 Aug 1;18(3):326-337. doi: 10.1016/j.cbpra.2010.09.001. PMID 21731410